CLINICAL TRIAL: NCT00410930
Title: Double-Blind Placebo-Controlled Study of Subcutaneous Immunotherapy in Birch Pollen Allergic Patients
Brief Title: Efficacy and Safety of Subcutaneous Immunotherapy in Birch Pollen Allergic Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DV08.01
Record Dates: First submitted 2006-12-12; First posted 2006-12-13 (Estimated); Last update posted 2006-12-19 (Estimated); Status verified 2006-12

CONDITIONS: Allergy
Keywords: Immunotherapy, major allergen, birch
MeSH Terms: conditions — Hypersensitivity

INTERVENTIONS:
Biological: Subcutaneous immunotherapy - Recombinant birch pollen

SUMMARY:
To compare versus placebo the efficacy and safety of recombinant Bet v1, natural purified Bet v1 and birch pollen licenced extract used for subcutaneous immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-50 with seasonal rhinoconjunctivitis for at least 2 years, and/or mild asthma range 1 and 2 GINA.
* Positive history of birch pollen allergy (clinical history, positive skin prick test, birch specific IgE, presence of birch pollen)
* Compliant patients
* Written consent.

Exclusion Criteria:

* Perennial rhinoconjunctivitis and/or asthma due to cosensitization with: animal danders, mites, alternaria cladosporium
* Uncontrolled seasonal asthma : severe asthma permanent or not range 3 and 4 of GINA.
* Patients treated with beta-blockers or under continuous oral corticosteroids.
* Pregnant women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160
Dates: Start 2002-11; Study Completion 2005-11

PRIMARY OUTCOMES:
Reduction of symptom and medication scores.

CONTACTS AND LOCATIONS:
Overall Officials: Gabrielle PAULI, MD, Pr, Principal Investigator — Hôpital Liautey - Strasbourg, France
Locations (1):
- Pr Gabrielle PAULI, Strasbourg, France